CLINICAL TRIAL: NCT03258502
Title: A Randomised, Phase 2a, Double-Blind, Placebo-Controlled Study To Evaluate The Safety, Pharmacokinetics And Antiviral Activity Of Multiple Doses Of RV521 Against Respiratory Syncytial Virus Infection In The Virus Challenge Model
Brief Title: A Study to Learn About the Effects of Multiple Doses of Sisunatovir on People With Respiratory Syncytial Virus (RSV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REVC002; C5241002 (Other: Alias Study Number)
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — sisunatovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RV521 (Experimental): RV521 drug substance in capsule for oral administration
  Interventions: Drug: RV521
- Placebo (Placebo Comparator): Micro-crystalline cellulose in capsule for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV521 — RV521 drug in capsules
  Arms: RV521
Drug: Placebo — Placebo in capsules
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn about the safety, pharmacokinetics and antiviral activity of the study medicine (called sisunatovir/RV521) for the potential treatment of respiratory syncytial virus (RSV). Sisunatovir will be given as multiple doses during the treatment period. RSV is a highly contagious virus that can lead to serious lung infections in patients with reduced ability to fight infection. Most vulnerable populations include babies, the elderly and patients that have received a bone marrow transplant.

This study is seeking healthy participants who are:

1. Aged 18 to 45 years old and will agree to the use of highly effective methods of contraception.
2. with a body mass index (BMI) of 18.0 to 30.0 Kg/m2 This study will consist of 2 cohorts of 33 participants each. In both cohorts participants will be exposed to the challenge virus on study day 0. Cohort 1 will receive either 200 mg of sisunatovir or placebo (looks the same as sisunatovir but contains no active medicine) 2 times a day for 5 days. Cohort 2 will receive either 350 mg of sisunatovir or placebo 2 times a day for 5 days. Participants will start taking the study medicine upon confirmation of RSV infection (or evening of Day 5 if not positive to RSV). The study medicine will be administered 12 hours apart (or twice daily). Each participant will remain in the quarantine unit until discharge on Day 12.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive
* In good health with no history of major medical conditions
* A total body weight ≥ 50 kg and a body mass index (BMI) of >/=18kg/m2 and </=30kg/m2

Exclusion Criteria:

* Evidence of any clinically significant or currently active major medical condition
* Positive for Human Immunodeficiency Virus, active Hepatitis A, B or C test
* Significant nose or nasopharynx abnormalities
* Abnormal lung function
* History or currently active symptoms suggestive of upper or lower respiratory tract infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in viral load | Baseline to study day 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- hVIVO Services Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] DeVincenzo J, Tait D, Efthimiou J, Mori J, Kim YI, Thomas E, Wilson L, Harland R, Mathews N, Cockerill S, Powell K, Littler E. A Randomized, Placebo-Controlled, Respiratory Syncytial Virus Human Challenge Study of the Antiviral Efficacy, Safety, and Pharmacokinetics of RV521, an Inhibitor of the RSV-F Protein. Antimicrob Agents Chemother. 2020 Jan 27;64(2):e01884-19. doi: 10.1128/AAC.01884-19. Print 2020 Jan 27. PMID 31712214
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=REVC002